CLINICAL TRIAL: NCT02200601
Title: Pre-Market Algorithm Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Force Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEIPHER_CLIN_002
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Seipher Wellness; algorithm; secure samples of SGC waveform; volunteers; validation; heart health algorithm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seipher Wellness (Experimental)
  Interventions: Device: Seipher Wellness

INTERVENTIONS:
Device: Seipher Wellness

SUMMARY:
The study sponsor has developed a patented medical device called Seipher Wellness. This is a non-invasive medical device that assesses heart health based on established cardiac parameters; timing events of the cardiac cycle. These are specific parameters captured and analyzed by the device. A ratio of two specific timing parameters provides an assessment of the subject's overall heart health. The aim of this study is to validate the device algorithm across a range of subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* able to understand the informed consent document
* willing to participate
* ambulatory volunteers

Exclusion Criteria:

* individuals with visible scar(s) or deformity in the test area of the chest
* non-ambulatory subjects
* enrolled in another concurrent study or trial
* exercised excessively within the last 4 hours
* unwilling to sign informed consent
* female subjects who are pregnant, suspected or planning to become pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Systolic Time Intervals (STI) value | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Houlton, MB ChB, Principal Investigator — Heart Force Medical
Locations (1):
- Integrative Naturopathic Medical Centre, Vancouver, British Columbia, Canada